CLINICAL TRIAL: NCT07031336
Title: Photon-counting CT Post-processing Protocols for Robust Quantifications in Chest CT Scans
Brief Title: Photon-counting CT in Chest Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00117084
Record Dates: First submitted 2025-06-02; First posted 2025-06-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Energy-integrating and photon-counting CT scans (Other): The participants will receive an energy-integrating CT scan as part of the main study (NCT00608764) and a photon-counting CT scan as part of this protocol.
  Interventions: Device: Photon-counting CT; Device: Energy-integrating CT

INTERVENTIONS:
Device: Photon-counting CT — The participants will receive a photon-counting CT scan as part of this protocol.
Device: Energy-integrating CT — The participants will receive an energy-integrating CT scan as part of the main study (NCT00608764).

SUMMARY:
Purpose and objective: This project aims to evaluate photon-counting computed tomography (PCCT) quantitative accuracy using COPDGene subjects. The goal is to establish acquisition protocols for PCCT scans with proper post-processing (e.g., reconstruction parameters and harmonization techniques) that enable reproducible measurements of emphysema metrics (e.g., Perc15, LAA-950, HU accuracy) and airways (Pi10, WA%) in the lungs.

Study activities and population group: The study will recruit subjects from a current study at Duke (COPDGene Phase 4, Pro00113442). Here are the aims:

* The research team will request consent from participants to acquire PCCT scans at their Phase 4 COPDGene visit. Scans will be performed using a PCCT-specific protocol.
* Reconstruct the PCCT images with multiple post-acquisition parameter settings. Apply harmonization techniques that are recently developed by the investigators of this study.

Data analysis:

* Identify the reconstruction and harmonization conditions that enable reproducible measurements of emphysema metrics (perc15, LAA-950, HU accuracy) and airways (Pi10, WA%), when compared to the counterpart EICT scans.
* Demonstrate the non-inferiority and potentially improved capabilities of PCCT scans in cross-sectional and longitudinal studies.

Risk/safety issues:

The participants are asked to get an additional CT scan with a PCCT scanner at their COPDGene Phase 4 visit. This additional CT scan will be done using an inspiratory chest protocol with a total of 3 mGy (~1.5 mSv) radiation dose. This is roughly equivalent of 6 month of background radiation. Women who are pregnant will not have a chest CT scan done until they are confirmed to be not pregnant.

ELIGIBILITY:
Inclusion Criteria:

* This study recruit from the Duke-COPDGene Phase 4 study. All participants from this cohort is eligible and they will be included if they consent.

Exclusion Criteria:

* This study recruit from the Duke-COPDGene Phase 4 study. All participants from this cohort is eligible and they will be included if they consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative reproducibility as measured by consistency of Perc15 (15th Percentile of lung CT histogram in Hounsfield Unit) | Day of Study Visit, approximately 30 minutes
  Perc15 will be measured from CT images, and its reproducibility will be quantified. The reproducibility of the measurements is defined as the least significant difference between two consecutive measurements across imaging conditions using the within-subject standard deviation method. The 95% confidence interval for reproducibility will be generated using a bootstrapping method with 5000 samples.
Quantitative reproducibility as measured by consistency of LAA-950 (Percentage of CT lung voxels below -950 Hounsfield Units) | Day of Study Visit, approximately 30 minutes
  LAA-950 will be measured from CT images, and its reproducibility will be quantified. The reproducibility of the measurements is defined as the least significant difference between two consecutive measurements across imaging conditions using the within-subject standard deviation method. The 95% confidence interval for reproducibility will be generated using a bootstrapping method with 5000 samples.
Quantitative reproducibility as measured by consistency of WA% (proportion of the airway wall area to the total airway area) | Day of Study Visit, approximately 30 minutes
  WA% will be measured from CT images, and its reproducibility will be quantified. The reproducibility of the measurements is defined as the least significant difference between two consecutive measurements across imaging conditions using the within-subject standard deviation method. The 95% confidence interval for reproducibility will be generated using a bootstrapping method with 5000 samples.
Quantitative reproducibility as measured by consistency of Pi10 (square root of airway wall area for a hypothetical airway with a 10 mm lumen perimeter) | Day of Study Visit, approximately 30 minutes
  Pi10 will be measured from CT images, and its reproducibility will be quantified. The reproducibility of the measurements is defined as the least significant difference between two consecutive measurements across imaging conditions using the within-subject standard deviation method. The 95% confidence interval for reproducibility will be generated using a bootstrapping method with 5000 samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Abadi, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No